CLINICAL TRIAL: NCT05001048
Title: Sex Differences in Sympathetic Activity and Vascular Reactivity During Acute and Chronic Hypoxia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00088122
Record Dates: First submitted 2021-08-04; First posted 2021-08-11 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Vasodilation; Vasoconstriction
MeSH Terms: conditions — Aneurysm | interventions — Phenylephrine

STUDY DESIGN:
Intervention Model Description: Participants will partake in all three arms of the study, which include: 1) low altitude, 2) early acclimatization, and 3) late acclimatization to high altitude assessments.
Masking Description: Due to the study design, masking is not possible. The time points and dosages of the study drug will be known to the participant. Further, due to the wash-out time of the acute hypoxia/hyperoxia interventions, these will always be completed second to the interventions breathing room air.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Altitude (Experimental): Participants will be assessed at an altitude of <1050m.
  Interventions: Drug: Phenylephrine Hydrochloride; Other: Cold Pressor Test; Other: Isocapnic Acute Hypoxia
- Early Acclimatization to High Altitude (Experimental): Participants will be assessed on day 2 or 3 of a high-altitude expedition at 3,800m.
  Interventions: Drug: Phenylephrine Hydrochloride; Other: Cold Pressor Test; Other: Hyperoxia
- Late Acclimatization to High Altitude (Experimental): Participants will be assessed on day 9 or 10 of a high-altitude expedition at 3,800m.
  Interventions: Drug: Phenylephrine Hydrochloride; Other: Cold Pressor Test; Other: Hyperoxia

INTERVENTIONS:
Drug: Phenylephrine Hydrochloride — Series of three incremental bolus injections to observe α1-adrenoreceptor mediated vasoconstriction.
  Other Names: Neo-Synephrine
Other: Cold Pressor Test — Standardized sympathetic stressor involving submersion of the hand in ice-cold water for 3-minutes, aiming to elicit endogenous neurotransmitter release and blood pressure increases.
Other: Isocapnic Acute Hypoxia — During low altitude assessment, participants will be exposed to isocapnic hypoxia equivalent to 3,800m to assess responses to acute exposure.
  Arms: Low Altitude
Other: Hyperoxia — During high altitude assessments, participants will breathe an oxygen concentration comparable to their end-tidal values at low altitude for the assessment of the influences of acclimatization.
  Arms: Early Acclimatization to High Altitude; Late Acclimatization to High Altitude

SUMMARY:
This study aims to investigate sex differences in blood pressure control associated with exposure to acute hypoxia (low oxygen), and short term acclimatization to hypoxia at high altitude.

DETAILED DESCRIPTION:
About 200 million people worldwide live at high altitudes. Millions of others travel to high altitude every year for work or travel. The low oxygen (or hypoxia) experienced at high altitudes causes considerable physiological stress, and the body adapts in order to maintain adequate oxygen delivery to its tissues. One of these adaptations is an increase in the activity of the sympathetic nervous system. This system is responsible for the "fight or flight" response. Sympathetic activity regulates the size of the blood vessels, which will affect blood pressure. Previous studies suggest that males and females regulate their blood pressure in different ways. Females tend to have lower resting sympathetic activity, and less vasoconstriction in response to stressors than males. Blood pressure changes are also influenced by levels of sex hormones; for example, estrogen may cause opposing vasodilation. Therefore, it is important to understand the differences in how males and females respond to low oxygen.

The main purpose of this study is to examine the differences between males and females in control of blood vessels during exposure to low oxygen. To study this question, we will test vasoreactivity to set physiological stressors in both males and females. Participants will be recruited at the Canadian sites, and we will test them while they breathe low oxygen for a short amount of time at low altitude. We will also perform assessments on the same participants during a two week stay at high altitude at White Mountain, CA, which is at an altitude of 3,800m. These data will have implications in the basic understanding of differences between male and female physiology. Specifically, to males and females living or travelling to high altitude.

ELIGIBILITY:
Inclusion Criteria:

* Between ages of 18-50
* No medical history of cardiovascular, respiratory, nervous system, or metabolic disease
* Females must be pre-menopausal

Exclusion Criteria:

* Any known cardiovascular, respiratory, nervous system, or metabolic disease (however, participants with controlled arterial hypertension will not be excluded)
* Having travelled above 2,000m within 1 month of testing at low and high altitude
* Females who are pregnant, confirmed by a pregnancy test
* Females who are post-menopausal
* Participants that are classified as obese (body mass index > 30kg⋅m²)
* Have a history of smoking regularly in the last 6 months (but nicotine substitutes (patch, gum) not an exclusion criteria)
* Those with a known allergy to sulfites
* Participants taking monoamine oxidase (MAO) inhibitors or tricyclic antidepressants

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-08-04 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | 18 minutes
  Phenylephrine sensitivity
Change in arterial blood flow | 18 minutes
  Phenylephrine sensitivity
Cold pressor test reactivity | 4 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Sean van Diepen, MD, MSc, Principal Investigator — University of Alberta; Craig Steinback, PhD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Mount Royal University, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta

REFERENCES:
- [Background] Hart EC, Charkoudian N, Wallin BG, Curry TB, Eisenach JH, Joyner MJ. Sex differences in sympathetic neural-hemodynamic balance: implications for human blood pressure regulation. Hypertension. 2009 Mar;53(3):571-6. doi: 10.1161/HYPERTENSIONAHA.108.126391. Epub 2009 Jan 26. PMID 19171792
- [Background] Mazzeo RS, Child A, Butterfield GE, Mawson JT, Zamudio S, Moore LG. Catecholamine response during 12 days of high-altitude exposure (4, 300 m) in women. J Appl Physiol (1985). 1998 Apr;84(4):1151-7. doi: 10.1152/jappl.1998.84.4.1151. PMID 9516178
- [Background] Purdy GM, James MA, Rees JL, Ondrus P, Keess JL, Day TA, Steinback CD. Spleen reactivity during incremental ascent to altitude. J Appl Physiol (1985). 2019 Jan 1;126(1):152-159. doi: 10.1152/japplphysiol.00753.2018. Epub 2018 Nov 21. PMID 30462566
- [Background] Usselman CW, Gimon TI, Nielson CA, Luchyshyn TA, Coverdale NS, Van Uum SH, Shoemaker JK. Menstrual cycle and sex effects on sympathetic responses to acute chemoreflex stress. Am J Physiol Heart Circ Physiol. 2015 Mar 15;308(6):H664-71. doi: 10.1152/ajpheart.00345.2014. Epub 2014 Dec 19. PMID 25527774